CLINICAL TRIAL: NCT03501966
Title: Randomized Trial of Medical Therapy (MT) vs. MT Plus Optic Nerve Sheath Fenestration vs. MT Plus Ventriculoperitoneal Cerebrospinal Fluid Shunting in Subjects With Idiopathic Intracranial Hypertension and Moderate to Severe Visual Loss
Brief Title: Surgical Idiopathic Intracranial Hypertension Treatment Trial
Acronym: SIGHT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH); University of Iowa (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIGHT; 1U10EY025990-01A1 (NIH)
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Results first posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2020-02

CONDITIONS: Idiopathic Intracranial Hypertension
Keywords: headache; idiopathic intracranial hypertension (IIH); shunt; fenestration; acetazolamide; visual loss; diamox
MeSH Terms: conditions — Pseudotumor Cerebri; Headache; Vision Disorders | interventions — Acetazolamide; Water; Diuretics

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned with equal allocation to one of the three treatment groups. Using a permuted block design, randomization will be stratified by PMD (average of 2 size V stimulus tests) in the eligible eye(s) (-6 dB to >-12 dB; -12 dB to >-20 dB; -20 dB to -27 dB). If a subject has two eligible eyes, the average PMD of the two eyes will be used for stratification.
Who Masked: Outcomes Assessor
Masking Description: Partially-masked technicians for perimetry, fundus photos, OCT, and refraction/ visual acuity
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Acetazolamide including Diet (Active Comparator): Subjects will use 250 mg tablets of acetazolamide, divided into two doses, taken with meals. Initial dose will be 1,000 mg twice per day and increased per titration schedule (Table 6 in protocol).
  Dietary consultation will include advising subjects to adopt a low sodium weight reduced diet.
  Interventions: Drug: Acetazolamide
- Optic Nerve Sheath Fenestration (Active Comparator): Acetazolamide including Diet plus Optic Nerve Sheath Fenestration (ONSF) Subjects will use 250 mg tablets of acetazolamide, divided into two doses, taken with meals. Initial dose will be 1,000 mg twice per day and increased per titration schedule (Table 6 in protocol).
  Dietary consultation will include advising subjects to adopt a low sodium weight reduced diet.
  ONSF performed by qualified, certified orbital surgeon using either a medial or supero-medial lid crease approach. ONSF will be performed in one or both eyes, depending on criteria.
  Interventions: Procedure: Optic Nerve Sheath Fenestration
- Ventriculoperitoneal CSF Shunting (Active Comparator): Acetazolamide including Diet plus Ventriculoperitoneal CSF Shunting (VPS) Subjects will use 250 mg tablets of acetazolamide, divided into two doses, taken with meals. Initial dose will be 1,000 mg twice per day and increased per titration schedule (Table 6 in protocol).
  Dietary consultation will include advising subjects to adopt a low sodium weight reduced diet.
  VPS performed by qualified, certified neurosurgeon using a frameless image-guided stereotactic system and positioning a shunt catheter in the lateral ventricle of the cerebral hemisphere not associated with speech. The catheter will be connected to an adjustable valve, and a distal shunt system will be placed in the peritoneal cavity.
  Interventions: Procedure: Ventriculoperitoneal CSF Shunting

INTERVENTIONS:
Drug: Acetazolamide — Medical therapy including diet
  Other Names: Diamox; water pill; diuretic
  Arms: Acetazolamide including Diet
Procedure: Optic Nerve Sheath Fenestration — Medical therapy including diet + optic nerve sheath fenestration
  Other Names: ONSF
  Arms: Optic Nerve Sheath Fenestration
Procedure: Ventriculoperitoneal CSF Shunting — Medical therapy including diet + ventriculoperitoneal CSF Shunting
  Other Names: VPS; CSF Shunt Surgery
  Arms: Ventriculoperitoneal CSF Shunting

SUMMARY:
Randomized trial of adults (≥18 years old) with idiopathic intracranial hypertension and moderate to severe visual loss without substantial recent treatment who are randomly assigned to (1) medical therapy, (2) medical therapy plus ONSF, or (3) medical therapy plus VPS. The primary outcome is visual field mean deviation change at first of Month 6 (26 weeks) or time of treatment failure of the eligible eye(s), followed by a continuation study to assess time to treatment failure. The determination of eligible eye(s) is based on meeting the eligibility criteria at baseline.

DETAILED DESCRIPTION:
After signing the informed consent form, potential subjects will be assessed for eligibility, including eliciting medical and neurologic history, measurement of best-corrected visual acuity, visual field testing, ophthalmoscopy with optic disc edema grading, physical examination, and Optical Coherence Tomography (OCT). Questionnaires will be completed. Blood will be drawn for complete blood count (CBC), electrolytes, liver function tests, renal function tests, amylase if not done as part of routine care within 4 weeks and a pregnancy test will be performed (women of childbearing potential).

Two visual field examinations using a size V stimulus will need to be performed at the Screening/Baseline Visit. The size V fields will be sent to the Visual Field Reading Center (VFRC) to confirm eligibility or determine that testing must be repeated for the subject.

Eligible individuals will be randomly assigned with equal allocation to one of 3 treatment groups: (1) medical therapy, (2) medical therapy plus ONSF, or (3) medical therapy plus VPS. Acetazolamide should be started on the day of randomization. Surgery should be performed as soon as possible, ideally within 3 days of randomization, but not more than 7 days.

Medical therapy will consist of a low sodium weight loss diet and acetazolamide with or without furosemide. Treatment will start with acetazolamide 2 grams per day, with the dose increased as tolerated up to 4 grams per day. If there is no clinical improvement after 2 weeks of maximal dosage of acetazolamide, furosemide will be started at a dose of 40 mg per day (along with potassium) and titrated up to 160-200 mg per day. Pharmacotherapy will be tapered when there is improvement in the papilledema grade, substantial improvement in the PMD and improvement in symptoms or when there is a safety concern.

The primary outcome is measured at the first of 6 months (26 weeks) or time of treatment failure. During the randomized trial, follow-up visits will occur after weeks 4, 8, 16, and 26 (± 7 days). Safety visits will occur after weeks 1 and 2 (± 4 days). Additional office visits may occur as needed. Phone contacts will occur at 12 and 20 weeks (±7 days).

After the 6-month primary outcome visit, subjects will transition to the Treatment Failure Identification Phase for up to 3 years. Ongoing treatment will continue following the guidelines for the first six months as long as treatment failure criteria are not met at which time treatment will be at the discretion of the Site Investigator. Investigators are urged to employ treatments from another arm of the study before other treatments under these circumstances.

ELIGIBILITY:
Inclusion Criteria:

* Subject Eligibility Criteria Inclusion Criteria

  1. Diagnosis of IIH by modified Dandy criteria (Table 4)
  2. Age 18 to <64 years at time of consent
  3. Age 18 to <61 years at time of diagnosis (time of diagnosis is the time at which the patient meets the modified Dandy criteria, usually after the lumbar puncture results are reviewed)
  4. Presence of bilateral papilledema
  5. Lumbar puncture within 6 weeks of screening visit or completed as part of screening: Opening CSF pressure >250 mmH2O or 200 to 250 mmH2O with at least one of the following:

     * Pulse synchronous tinnitus
     * Cranial nerve VI palsy
     * Echography for disc drusen negative and no other disc anomalies mimicking disc edema present
     * Magnetic Resonance Venography (MRV) with lateral sinus collapse/stenosis, partially empty sella turcica on coronal or sagittal views of MRI, and optic nerve sheaths with filled out CSF spaces next to the globe on T2 weighted axial MRI scans If the patient was treated with intracranial pressure lowering agents (e.g., acetazolamide) prior to obtaining a lumbar puncture, the agent(s) must be discontinued for at least 24 hours prior to performing the diagnostic lumbar puncture.
  6. At least one eye meeting all eligible eye inclusion criteria and no exclusion criteria.
  7. Able to provide informed consent
  8. Investigator believes participant is a good candidate for the study, including the probability of returning for follow-up.
* Eye-Level Eligibility Criteria Subjects must have at least one eye meeting all of the inclusion criteria and none of the exclusion criteria.

If both eyes meet eligibility criteria at the baseline examination, both will be included in the primary outcome analysis.

Inclusion

1. Visual field loss meeting the following criteria based on two full threshold 24-2 size V tests reviewed by the VFRC:

   * PMD from -6 decibel (dB) to -27 dB
   * Reproducible visual loss present on automated perimetry including no more than 15% false positive response
2. Visual acuity better than 20/200 (39 or more letters correct)

Exclusion Criteria:

* Subject Exclusion Criteria Exclusion Criteria

  1. Treatment of IIH within the past 3 months with either (1) the maximally tolerated dosage of acetazolamide for at least one week or (2) more than one month of acetazolamide with a cumulative dosage of more than 45 grams 'Maximally-tolerated dose' is defined as dosage was reached where dosage could not be increased further either because of side effects or because a daily total dosage of 4 grams per day was reached.

     If individual discontinued acetazolamide in the past due to side effects, individual is only eligible if investigator believes that the individual is likely to tolerate acetazolamide, as it will be prescribed in the study.
  2. Treatment of IIH within the past 3 months with either (1) the maximally tolerated dosage of methazolamide for at least one week or (2) more than one month of methazolamide with a cumulative dosage of more than 4.5 grams 'Maximally-tolerated dose' is defined as dosage was reached where dosage could not be increased further either because of side effects or because a daily total dosage of 400 mg per day was reached.
  3. Treatment with topiramate within two months and average cumulative dosage for the preceding month of more than 700 mg per week
  4. Previous surgery for IIH, including ONSF, CSF shunting, subtemporal decompression, or venous sinus stenting; gastric surgery for obesity is allowed
  5. Abnormalities on neurologic examination except for papilledema and its related visual loss or cranial nerve VI to VII paresis; if other abnormalities are present, the patient will need to be discussed with the Study Director (SD) for study entry.
  6. Abnormal CT or MRI scan (intracranial mass, hydrocephalus, dural sinus thrombus, or arteriovenous malformation) other than findings known to occur with increased intracranial pressure. Abnormalities on MRI that are not known to cause increased intracranial pressure are acceptable.
  7. Abnormal CSF contents: increased cells: > 8 cells; elevated protein: > 45 mg%; low glucose: < 30 mg% (If the lumbar puncture produces a cell count compatible with a traumatic needle insertion, the patient does not need to be excluded if the CSF white blood cell count (WBC) after correction is 8 cells/mm3 or less - see Manual of Procedures (MOP) for calculation. If > 8 cells or > 45mg% in CSF protein are documented in the CSF or calculated after conversion from a traumatic lumbar puncture, the patient can be discussed with the Study Director for possible inclusion.)
  8. Abnormal blood work-up indicating a medical or systemic condition associated with raised intracranial pressure
  9. Diabetes mellitus with diabetic retinopathy
  10. Ingestion of a drug or substance, or presence of a disorder, that has been associated with increased intracranial pressure within 2 months of diagnosis, such as lithium, vitamin A related products (e.g., Retin-A), or various cyclines (see MOP for conditions and drugs)
  11. Laboratory test results showing severe anemia, leukopenia or thrombocytopenia, renal failure, or hepatic disease, based on the Site Investigator's judgment
  12. Other condition requiring continued use of oral, I.V. or injectable steroids (nasal, inhaled, or topical steroids are allowed since the systemic effects are small). Patients with a condition that resulted in recent or current use of steroids but may be safely tapered off will be handled on a case-by-case basis after discussion with Study Director/co-Director. See Manual of Procedures (MOP) for details.
  13. Presence of a medical condition that would contraindicate use of acetazolamide or furosemide or significantly increase surgical risk
  14. Pregnancy or unwillingness for a subject of childbearing potential to use contraception during the first 6 months of the study Women of childbearing potential must use an acceptable form of birth control during the first 6 months of the study. Acceptable forms include oral contraceptives, transdermal contraceptives, diaphragm, intrauterine devices (IUDs), condoms with spermicide, documented surgical sterilization of either the subject or their partner, or abstinence.
  15. Presence of a physical, mental, or social condition likely to affect follow-up (drug addiction, terminal illness, no telephone, homeless)
  16. Anticipation of a move from the site area within six months and unwillingness to return for follow-up at a SIGHT study site
  17. Allergy to pupil dilating drops or narrow angles precluding safe dilation
  18. Presence of a condition that contraindicates general anesthesia
  19. Participation in an investigational trial within 30 days of enrollment that involved treatment with any systemic drug therapy or therapy that affects the eligible eye(s)
* Eye Level Exclusion Criteria Exclusion

  1. Intraocular pressure currently >28 mm Hg or >30 mm Hg at any time in the past
  2. Refractive error of more than -6.00 or more than +6.00 sphere or more than 3.00 cylinder with the following exceptions:

     * Eyes with more than 6.00 D of myopia but less than 8.00 D of myopia are eligible if: 1) there are no abnormalities on ophthalmoscopy related to myopia that are associated with visual loss (such as staphyloma, retinal thinning in the posterior pole, or more than mild optic disc tilt), and 2) the individual will wear a contact lens for all perimetry examinations with the appropriate correction.
     * Eyes with more than 6.00 D of hyperopia but less than 8.00 D of hyperopia are eligible if: 1) there is an unambiguous characteristic halo of peripapillary edema as opposed to features of a small crowded disc or other hyperopic change related to visual loss determined by the Site Investigator or the Photographic Reading Center (PRC) Director (or his designate), and 2) the individual will wear a contact lens for all perimetry examinations with the appropriate correction (which can be corrected for perimetry or with the patient's own contact lens with over correction by lens at the perimeter).

     Note: Refractive error exclusion and exceptions refer to sphere not spherical equivalent, with cylinder expressed in plus format.
  3. Other disorders causing visual loss except for refractive error and amblyopia, including cells in the vitreous or iritis
  4. Large optic disc drusen on exam or known in previous history (small drusen of the disc can occur with longstanding papilledema and are allowed if not so numerous that investigator determines they are contributing to vision loss)

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wall, MD, Study Director — University of Iowa
Locations (36):
- United States (33):
  - University of Southern California, Los Angeles, California
  - NeuroEyeOrbit Institute, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of Colorado - Anschutz Medical Campus, Aurora, Colorado
  - The Eye Care Group, Orange, Connecticut
  - University of Miami, Miami, Florida
  - Northwestern Medicine, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas School of Medicine, Prairie Village, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Bethesda Neurology, LLC, North Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Saint Louis University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - State University of New York at Stony Brook, East Setauket, New York
  - New York Eye & Ear Infirmary of Mount Sinai, New York, New York
  - New York University School of Medicine, New York, New York
  - University of Rochester, Rochester, New York
  - Ohio Neuro-Ophthalmology, Orbital Disease and Oculoplastics, Columbus, Ohio
  - Dean McGee Eye Institute, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Neuro-Eye Clinical Trials-Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Sunnybrook Health Science Center, Toronto, Ontario
- Rivera, Enrique J, Bayamón, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in October 2018 and continued until the study stopped on August 28, 2019.
Groups:
- Acetazolamide Including Diet: Subjects will use 250 mg tablets of acetazolamide, divided into two doses, taken with meals. Initial dose will be 1,000 mg twice per day and increased per titration schedule (Table 6 in protocol).
  Dietary consultation will include advising subjects to adopt a low sodium weight reduced diet.
  Acetazolamide: Medical therapy including diet
- Optic Nerve Sheath Fenestration: Acetazolamide including Diet plus Optic Nerve Sheath Fenestration (ONSF) Subjects will use 250 mg tablets of acetazolamide, divided into two doses, taken with meals. Initial dose will be 1,000 mg twice per day and increased per titration schedule (Table 6 in protocol).
  Dietary consultation will include advising subjects to adopt a low sodium weight reduced diet.
  ONSF performed by qualified, certified orbital surgeon using either a medial or supero-medial lid crease approach. ONSF will be performed in one or both eyes, depending on criteria.
  Optic Nerve Sheath Fenestration: Medical therapy including diet + optic nerve sheath fenestration
- Ventriculoperitoneal CSF Shunting: Acetazolamide including Diet plus Ventriculoperitoneal CSF Shunting (VPS) Subjects will use 250 mg tablets of acetazolamide, divided into two doses, taken with meals. Initial dose will be 1,000 mg twice per day and increased per titration schedule (Table 6 in protocol).
  Dietary consultation will include advising subjects to adopt a low sodium weight reduced diet.
  VPS performed by qualified, certified neurosurgeon using a frameless image-guided stereotactic system and positioning a shunt catheter in the lateral ventricle of the cerebral hemisphere not associated with speech. The catheter will be connected to an adjustable valve, and a distal shunt system will be placed in the peritoneal cavity.
  Ventriculoperitoneal CSF Shunting: Medical therapy including diet + ventriculoperitoneal CSF Shunting
Period: Overall Study
Arm/Group | Acetazolamide Including Diet | Optic Nerve Sheath Fenestration | Ventriculoperitoneal CSF Shunting
Started | 2 | 2 | 3
Completed | 0 | 0 | 0
Not Completed | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Population: No data collected, study terminated due to poor enrollment prior to any data collection.
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetazolamide Including Diet | Optic Nerve Sheath Fenestration | Ventriculoperitoneal CSF Shunting | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Perimetric Mean Deviation (PMD)
Description: Change from baseline to first of Month 6 (Week 26) or time of treatment failure in PMD (perimetric mean deviation) in eligible eye(s) with the size V stimulus
Time Frame: 6 months
Population: No data collected, study terminated due to poor enrollment prior to any data collection.
Arm/Group | Acetazolamide Including Diet | Optic Nerve Sheath Fenestration | Ventriculoperitoneal CSF Shunting
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Treatment Failure
Description: Time from randomization to treatment failure
Time Frame: up to 3 years
Population: No data collected, study terminated due to poor enrollment prior to any data collection.
Arm/Group | Acetazolamide Including Diet | Optic Nerve Sheath Fenestration | Ventriculoperitoneal CSF Shunting
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Cerebrospinal Fluid (CSF) Opening Pressure
Description: Change in CSF opening pressure measurement by lumbar puncture
Time Frame: 6 months
Population: No data collected, study terminated due to poor enrollment prior to any data collection.
Arm/Group | Acetazolamide Including Diet | Optic Nerve Sheath Fenestration | Ventriculoperitoneal CSF Shunting
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Papilledema Grade
Description: Change in papilledema grade
Time Frame: 6 months
Population: No data collected, study terminated due to poor enrollment prior to any data collection.
Arm/Group | Acetazolamide Including Diet | Optic Nerve Sheath Fenestration | Ventriculoperitoneal CSF Shunting
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: OCT Retinal Nerve Fiber Layer Thickness
Description: Change in retinal nerve fiber layer thickness
Time Frame: 6 months
Population: No data collected, study terminated due to poor enrollment prior to any data collection.
Arm/Group | Acetazolamide Including Diet | Optic Nerve Sheath Fenestration | Ventriculoperitoneal CSF Shunting
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: OCT Total Retinal Thickness
Description: Change in total retinal thickness
Time Frame: 6 months
Population: No data collected, study terminated due to poor enrollment prior to any data collection.
Arm/Group | Acetazolamide Including Diet | Optic Nerve Sheath Fenestration | Ventriculoperitoneal CSF Shunting
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Visual Acuity (VA) Using Early Treatment Diabetic Retinopathy Study (ETDRS) Chart
Description: Change in VA scores, determined by baseline VA of better than 20/200 (39 or more letters correct) and worsening indicated by less correct letters
Time Frame: 6 months
Population: No data collected, study terminated due to poor enrollment prior to any data collection.
Arm/Group | Acetazolamide Including Diet | Optic Nerve Sheath Fenestration | Ventriculoperitoneal CSF Shunting
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Quality of Life (QoL) 36 Item Short Form Health Survey (SF-36v2)
Description: Changes in QoL as measured by responses
Time Frame: 6 months
Population: No data collected, study terminated due to poor enrollment prior to any data collection.
Arm/Group | Acetazolamide Including Diet | Optic Nerve Sheath Fenestration | Ventriculoperitoneal CSF Shunting
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Quality of Life (QoL) Visual Function Questionnaire (VFQ-25)
Description: Changes in QoL as measured by responses
Time Frame: 6 months
Population: No data collected, study terminated due to poor enrollment prior to any data collection.
Arm/Group | Acetazolamide Including Diet | Optic Nerve Sheath Fenestration | Ventriculoperitoneal CSF Shunting
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Quality of Life (QoL) 10-item Neuro-ophthalmic Supplement to the VFQ-25
Description: Changes in QoL as measured by responses
Time Frame: 6 months
Population: No data collected, study terminated due to poor enrollment prior to any data collection.
Arm/Group | Acetazolamide Including Diet | Optic Nerve Sheath Fenestration | Ventriculoperitoneal CSF Shunting
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Acetazolamide Including Diet | Optic Nerve Sheath Fenestration | Ventriculoperitoneal CSF Shunting
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT03501966/Prot_001.pdf
  • Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/66/NCT03501966/SAP_002.pdf
  • Informed Consent Form (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT03501966/ICF_000.pdf